CLINICAL TRIAL: NCT04491175
Title: Addressing Opioid Use Disorder With an External Multimodal Neuromodulation Device: Development and Clinical Evaluation of DuoTherm for Opioid-Sparing Pain Relief in Acute and Chronic Low Back Pain
Brief Title: Impact of DuoTherm on Opioid Use and Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MMJ Labs LLC (Industry)
Collaborators: Sport and Spine Rehab Clinical Research Foundation (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Amy Lynn Baxter, CEO, MMJ Labs LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Duotherm; 4R44DA049631-02 (NIH); R44DA058952 (NIH)
Record Dates: First submitted 2019-09-15; First posted 2020-07-29 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use; Low Back Pain
Keywords: chronic pain; analgesia; medical device; opioid; low back pain; neuromodulation; multifidus
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Agnosia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind controlled trial with 3- (aLBP) or 6- month (cLPB) follow-up.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants were blinded to which device powered the study hypothesis, and blinded to their assigned intervention until after documenting initial NRS pain intensity. The protocol statistician and study coordinator knew device assignments and had access to data, but did not conduct analysis. The PI and treating chiropractor were blinded to allocation and all data during enrollment, with the PI accessing data only after study completion. The analyzing statisticians were blinded to device assignment until completion of analysis. Success of participant blinding was tested with prompts, "select if you received… control or treatment" and "How confident are you?"
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Multimodal Harmonic Mechanical Stimulation Neuromodulation Wearable Belt (M-Stim) (Experimental): DuoTherm is a novel multimodal low back pain relief device incorporating 8 harmonic vibration patterns of mechanical stimulation (M-Stim) including neuromodulatory frequencies, 5 intensity levels, and optional heat, cold, and pressure delivered through a sculpted metal plate attached with a belt and controlled by buttons on the belt. Patients will be instructed to use the device at least daily for 30 minutes.
  Interventions: Device: M-Stim
- Transcutaneous Electrical Nerve Stimulation (TENS) (Active Comparator): A prescription 4-lead 8-channel TENS unit (LG Smart) with variable intensity settings. Patients will be instructed to use the TENS at least daily for 30 minutes.
  Interventions: Device: TENS

INTERVENTIONS:
Device: M-Stim — The casing for the device is a 54" belt with 3-button haptic controller for on-off, therapy cycles(8) and intensity(5) levels.
  Other Names: DuoTherm; Multiple VibraCool M-Stim units in a harmonic array on a thermoconductive plate with optional cold, heat, and pressure
  Arms: Multimodal Harmonic Mechanical Stimulation Neuromodulation Wearable Belt (M-Stim)
Device: TENS — LG SMART TENS stimulator is a portable electrotherapy devcie featuring transcutaneous electrical nerve stimulation (TENS) therapeutic device, which is used for pain relief. The stimulator sends a gentle electrical current to underlying nerves and muscle groups via electrodes applied on the skin. The parameters of the device are controlled by buttons on a controller with an adjustable intensity level.
  Other Names: LG Smart TENS
  Arms: Transcutaneous Electrical Nerve Stimulation (TENS)

SUMMARY:
Evaluate the difference in opioid use, pain intensity and pain interference in patients with moderate to severe low back pain using DuoTherm multimodal harmonic mechanical stimulation (M-Stim) unit compared to Transcutaneous Electrical Nerve Stimulation (TENS)

DETAILED DESCRIPTION:
160 patients with acute or exacerbations of chronic low back pain (LBP) presenting for chiropractic and rehabilitation care will be randomized to one of two conditions: an M-Stim pain relief belt device incorporating 8 patterns of vibration motors (and optional heat, cold, and pressure) delivered through a sculpted metal plate; or a 4-lead TENS unit with 8 channels of stimulation and adjustable intensity. Patients will be blinded to the hypothesis-driving intervention. They will be prompted daily by a Qualtrics text link to a secure data recording site collecting analgesic use and treatments, including opioid brand, dose, pill number, and source, and pain data, then weekly for 3 months (acute pain) or 6 months (chronic).

ELIGIBILITY:
Inclusion Criteria:

* Age18-90
* Moderate-to-severe low back pain with numeric rating scale >=4/10
* Capacity to understand informed consent
* Willingness to communicate prescriptions, pill number, dose, and source of opioids used

Exclusion Criteria:

* Opioid prescription in the past month for acute LBP (new pain <3 months)
* Radicular pain
* BMI greater than 50 (device won't fit)
* Sensitivity to cold or vibration (e.g Raynaud's or Sickle Cell Disease)
* Diabetic neuropathy
* New neurologic deficits
* Skin lesions over the low back area
* Contraindication to any medication for pain management
* Inability to apply DuoTherm or TENS device
* Pacemaker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Opioid initiation in the opioid-naive | All opioid diaries for 3 months
  New opioid prescriptions for subjects without history of opioids for LBP
Opioid use in prior users | 28 days (duration of daily recording)
  Change in milligram morphine equivalents (MME) reported daily

SECONDARY OUTCOMES:
Opioid Use Risk Factors in the Opioid-Naive | All opioid diaries for 3 months
  The difference in opioid use days, MME, and those using opioids more than 7 days after presentation
Opioid use in those with more severe pain | All opioid diaries for 6 months
  Opioid use days in those with the NIH Research Taskforce severity of moderate to severe in M-Stim versus TENS
Opioid prescribing compared to a contemporaneous national LPB prescribing of 25% | All opioid diaries for 6 months
  New opioid prescription rate for each intervention compared to nationally prevalent prescribing rates of 25% with moderate to severe pain in outpatient settings

CONTACTS AND LOCATIONS:
Overall Officials: Jena Slaski, Study Director — Sport and Spine Clinical Research Foundation
Locations (2):
- United States (2):
  - Sport and Spine Rehab Clinics, Landover, Maryland
  - Kaizo Health Fairfax, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the clinical results reported in any publications, after deidentification, will be available for a period of 36 months after publication to achieve approved aims of any researcher who provides a methodologically sound proposal. Proposals should be directed to info@mmjlabs.com. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: up to 36 months after publication of results
Access Criteria: researchers providing approved methodologically sound proposals

REFERENCES:
- [Background] Stumbo SP, Yarborough BJ, McCarty D, Weisner C, Green CA. Patient-reported pathways to opioid use disorders and pain-related barriers to treatment engagement. J Subst Abuse Treat. 2017 Feb;73:47-54. doi: 10.1016/j.jsat.2016.11.003. Epub 2016 Nov 15. PMID 28017184
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, Delitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. Phys Ther. 2015 Feb;95(2):e1-e18. doi: 10.2522/ptj.2015.95.2.e1. PMID 25639530
- [Background] Davis CS, Lieberman AJ, Hernandez-Delgado H, Suba C. Laws limiting the prescribing or dispensing of opioids for acute pain in the United States: A national systematic legal review. Drug Alcohol Depend. 2019 Jan 1;194:166-172. doi: 10.1016/j.drugalcdep.2018.09.022. Epub 2018 Nov 3. PMID 30445274
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Darnall BD, Colloca L. Optimizing Placebo and Minimizing Nocebo to Reduce Pain, Catastrophizing, and Opioid Use: A Review of the Science and an Evidence-Informed Clinical Toolkit. Int Rev Neurobiol. 2018;139:129-157. doi: 10.1016/bs.irn.2018.07.022. Epub 2018 Aug 6. PMID 30146045
- [Background] French SD, Cameron M, Walker BF, Reggars JW, Esterman AJ. Superficial heat or cold for low back pain. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD004750. doi: 10.1002/14651858.CD004750.pub2. PMID 16437495
- [Background] Farber K, Wieland LS. Massage for Low-back Pain. Explore (NY). 2016 May-Jun;12(3):215-7. doi: 10.1016/j.explore.2016.02.014. Epub 2016 Mar 2. PMID 27033320
- [Background] Nadler SF, Steiner DJ, Petty SR, Erasala GN, Hengehold DA, Weingand KW. Overnight use of continuous low-level heatwrap therapy for relief of low back pain. Arch Phys Med Rehabil. 2003 Mar;84(3):335-42. doi: 10.1053/apmr.2003.50103. PMID 12638100
- [Background] Delitto A, Patterson CG, Stevans JM, Freburger JK, Khoja SS, Schneider MJ, Greco CM, Freel JA, Sowa GA, Wasan AD, Brennan GP, Hunter SJ, Minick KI, Wegener ST, Ephraim PL, Beneciuk JM, George SZ, Saper RB. Stratified care to prevent chronic low back pain in high-risk patients: The TARGET trial. A multi-site pragmatic cluster randomized trial. EClinicalMedicine. 2021 Mar 30;34:100795. doi: 10.1016/j.eclinm.2021.100795. eCollection 2021 Apr. PMID 33870150
- [Background] Deyo RA, Hallvik SE, Hildebran C, Marino M, Dexter E, Irvine JM, O'Kane N, Van Otterloo J, Wright DA, Leichtling G, Millet LM. Association Between Initial Opioid Prescribing Patterns and Subsequent Long-Term Use Among Opioid-Naive Patients: A Statewide Retrospective Cohort Study. J Gen Intern Med. 2017 Jan;32(1):21-27. doi: 10.1007/s11606-016-3810-3. Epub 2016 Aug 2. PMID 27484682
- [Background] Hayden JA, Ellis J, Asbridge M, Ogilvie R, Merdad R, Grant DAG, Stewart SA, Campbell S. Prolonged opioid use among opioid-naive individuals after prescription for nonspecific low back pain in the emergency department. Pain. 2021 Mar 1;162(3):740-748. doi: 10.1097/j.pain.0000000000002075. PMID 32947539
- [Background] Baxter AL, Thrasher A, Etnoyer-Slaski JL, Cohen LL. Multimodal mechanical stimulation reduces acute and chronic low back pain: Pilot data from a HEAL phase 1 study. Front Pain Res (Lausanne). 2023 Apr 26;4:1114633. doi: 10.3389/fpain.2023.1114633. eCollection 2023. PMID 37179530
- [Derived] Baxter AL, Etnoyer-Slaski JL, Williams JAR, Swartout K, Cohen LL, Lawson ML. Preventing opioid prescribing for low back pain using multimodal mechanical stimulation vs. TENS: a randomized-controlled trial. Front Pain Res (Lausanne). 2025 Jul 10;6:1612572. doi: 10.3389/fpain.2025.1612572. eCollection 2025. PMID 40709052

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT04491175/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT04491175/ICF_000.pdf